CLINICAL TRIAL: NCT02326844
Title: A Phase 2 Pilot Study of BMN 673 (Talazoparib), an Oral PARP Inhibitor, in Patients With Deleterious BRCA1/2 Mutation-Associated Ovarian Cancer Who Have Had Prior PARP Inhibitor Treatment
Brief Title: BMN 673 (Talazoparib), an Oral PARP Inhibitor, in People With Deleterious BRCA1/2 Mutation-Associated Ovarian Cancer Who Have Had Prior PARP Inhibitor Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed by the Cancer Therapy Evaluation Program (CTEP)
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jung-Min Lee, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150050; 15-C-0050
Record Dates: First submitted 2014-12-25; First posted 2014-12-30 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Cancer
Keywords: Germline BRCA1/2 Mutations (gBRCAm); DNA Damaging Agents; FOX03a, 53BP1 and RAD51
MeSH Terms: conditions — Ovarian Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ovarian Cancer Patients (Experimental): Ovarian cancer patients with germline breast cancer mutation (gBRCAm) who have progressed on prior poly (ADP-ribose) polymerase inhibitor (PARPi) therapy
  Interventions: Drug: BMN 673 (talazoparib)

INTERVENTIONS:
Drug: BMN 673 (talazoparib) — 1 mg by mouth (p.o.) once daily on 28-day cycles until disease progression
  Other Names: talazoparib

SUMMARY:
Background:

- The new drug BMN 673 (talazoparib) has been shown to fight tumor cells in animals and some people. It is a poly (ADP-ribose) polymerase (PARP) inhibitor. It works on tumor cell deoxyribonucleic acid (DNA) damage repair process. Researchers want to see if BMN 673 shrinks cancer again in women with ovarian cancer and whose cancer initially got shrunk but grew back on the first PARP inhibitor.

Objective:

- To study BMN 673 (talazoparib) in people with ovarian cancer born with a breast cancer (BRCA) mutation and whose cancer got shrunk but became worse after they took a similar drug.

Eligibility:

* Women at least 18 years old:
* with recurrent and/or metastatic germline breast cancer mutation (gBRCAm)-associated ovarian cancer AND
* whose disease is growing after already being treated with PARP inhibitors AND
* with no other treatment(s) in between the first PARP inhibitors and a screening visit.

Design:

* Participants will be screened with medical history, physical exam, and heart and blood tests.
* Participants will take the study drug by mouth once daily. They will take the drug in 28-day cycles.
* They will keep a diary of doses and any side effects.
* Participants will have 4 study visits in cycle 1, then 1 visit every cycle. Visits may include:
* Blood tests
* Physical exam
* Computed tomography (CT) or magnetic resonance imaging (MRI) scans. Participants will lie in a machine that takes pictures of their body.
* Ultrasound
* Participants will have a biopsy before starting the study drug. A small piece of tumor tissue will be removed by needle, guided by a scan. They may have two more biopsies later.
* Participants will be followed for 30 days after taking the last dose of study drug. A physical exam, blood tests, and CT or other scans will be done.
* Participants will have follow-up calls to ask about any side effects.

DETAILED DESCRIPTION:
Background:

* Patients with germline BRCA1/2 mutations (gBRCAm) demonstrate repeated therapeutic susceptibility to deoxyribonucleic acid (DNA) damaging agents, especially platinums, even if they have previously progressed on a similar (platinum-based) regimen.
* Poly (ADP-ribose) polymerase (PARP) inhibitors (PARPi) have clinical activity in gBRCAm-associated malignancies, although patients eventually develop progressive disease.
* BMN 673 (talazoparib) is a novel PARPi, with excellent oral bioavailability and greater anti-tumor activity in vitro and in vivo at lower concentrations than first generation PARPi.
* It is unknown whether secondary BRCA mutations or other potential mechanisms of clinical resistance portend cross-resistance to a highly potent PARPi.

Objectives:

-To determine the objective response rate (complete response (CR)+partial response (PR)) of single agent BMN 673 (talazoparib) in ovarian cancer patients with gBRCAm who have progressed on prior PARPi therapy.

Eligibility:

* Women with recurrent and/or metastatic gBRCAm-associated ovarian cancer, with progression on PARPi monotherapy within the immediate prior 2 months of the time of screening visit.
* Patients should have responded to their prior PARPi therapy (CR, PR or stable disease (SD)>4months).
* Patients cannot have received another therapy between stopping their first PARPi therapy\ and initiating therapy on this trial, but must be off the prior PARPi for at least 4 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 and adequate organ and marrow function.

Design:

* This is an open label, single arm phase II trial to examine activity of BMN 673 (talazoparib).
* Patients will receive BMN 673 (talazoparib) at the recommended phase 2 dose (RP2D) of 1mg p.o. once daily on 28 day cycles.
* Research samples including whole blood, plasma, circulating tumor cells (CTCs), and tumor biopsies will be obtained for progressive disease (PD) endpoints at baseline, cycle 1 day 29 (prior to cycle 2 day 1), and/or at progression in all patients.
* Patients will be evaluated every two cycles for response using Response Evaluation Criteria in Solid Tumors (RECIST)v1.1 criteria and every cycle for safety using Common Terminology Criteria in Adverse Events (CTCAE)v4.0.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Recurrent, and/or metastatic germline breast cancer (BRCA) 1/2 mutation-associated ovarian cancer, with progression on a poly (ADP-ribose) polymerase (PARP) inhibitor monotherapy after attaining a response to that PARPi (complete response (CR), partial response (PR), or stable disease (SD) greater than or equal to 4mo)
* Progression should have occurred within the immediate prior 2 months of the time of screening visit, with no intervening anti-cancer therapy.
* Patients must be at least 4 weeks from the last dose of prior PARP inhibitor.
* All patients must have at least one lesion deemed safe to biopsy and be willing to undergo mandatory baseline biopsy. It is preferred that this lesion be a lesion that progressed or arose while on the prior PARP therapy.
* Histopathologic diagnosis of ovarian cancer (including primary peritoneal and fallopian tube cancers) must be confirmed in the Laboratory of Pathology, National Cancer Institute (NCI).
* Age greater than or equal to18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to100,000/mcL
  * total bilirubin less than or equal to 1.5X upper limit of normal, unless known Gilberts syndrome
  * Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 x institutional upper limit of normal
  * creatinine < 1.5 X upper limit of normal

OR

* measured creatinine clearance >60 mL/min/1.73 m(2) for patients with serum creatinine levels > 1.5 x upper limit of normal.
* hemoglobin greater than or equal to 10 mg/dL (in the absence of transfusion within 24 hours prior to dosing).

  * All patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST).
  * Use of raloxifene for bone health is allowed.
  * Patients must be at least 1 week from the last dose of complementary or alternative medications.
  * Patients who have had major surgery must be fully recovered and greater than or equal to 4 weeks postoperative prior to enrolling on study.
  * Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study

participation, and for at least three months following the last dose of experimental therapy and must have a negative urine or serum pregnancy test within 7 days prior to the start of the study.

* Patient must be able to swallow pills.
* Integral biomarkers: all patients who are eligible for the study due to a history of positive BRCA1/2 mutation must provide documented evidence of their deleterious germline mutation status, obtained in a Clinical Laboratory Improvement Amendment (CLIA)-certified laboratory, including but not limited to Myriad Genetics prior to study enrollment. Variants of uncertain significance (VUS) of BRCA1/2 and BRCA1/2 somatic mutations are not considered deleterious germline BRCA1/2 mutations. Due to the long acceptance of BRCA 1 and BRCA 2 mutation testing through Myriad, Myriad results will be acceptable. If testing for BRCA 1 and BRCA 2 mutation is done by other organizations, a genetic consultation report from a qualified medical professional confirming that the laboratory results showed a recognized germ line deleterious BRCA 1 or BRCA 2 mutation or deleterious BRCA 1 rearrangement is required.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had prior BMN 673 (talazoparib) therapy.
* Patients with known brain metastases diagnosed within 1 year will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Exception: patients with brain metastases diagnosed greater than 1 year prior to study entry may be considered if they received sterilizing therapy to the central nervous system (CNS) (resection or radiation) and have been CNS progression-free for the 1-year period.
* Lack of recovery of prior cancer therapy-related adverse events to Grade less than or equal to 1 (National Cancer Institute (NCI) Common Terminology Criteria in Adverse Events (CTCAE) v4.03; except alopecia). Stable persistent grade 2 peripheral neuropathy may be allowed as determined on a case-by-case basis at the discretion of the PI. Patients with platinum-related grade 2 or greater hypomagnesemia (on replacement) will be eligible.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, clinically significant gastrointestinal (GI) bleeding or hemoptysis within 28 days prior to the start of the study, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with active infection will not be eligible, but may become eligible once infection has resolved and they are at least 7 days from completion of antibiotics.
* Another previous or current invasive malignancy within the last 2 years, with the exception of curatively treated stage Ia cervical carcinoma, or resected stage Ia endometrial cancer, and noninvasive nonmelanoma skin cancers.
* Human immunodeficiency virus (HIV)- positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with BMN 673 (talazoparib). HIV- positive patients who are not on combination antiretroviral therapy (cART) and have cluster of differentiation 4 (CD4) counts > 500 are eligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BMN 673 (talazoparib)

Patients who are receiving any other investigational or commercial agents with the intent to treat the malignancy.

* Patients with gastrointestinal conditions that might predispose for drug intolerability or poor drug absorption.
* Use of nasogastric or gastric (G)-tube administration.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2016-04-14 (Actual); Study Completion 2016-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Min Lee, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JM, Hays JL, Annunziata CM, Noonan AM, Minasian L, Zujewski JA, Yu M, Gordon N, Ji J, Sissung TM, Figg WD, Azad N, Wood BJ, Doroshow J, Kohn EC. Phase I/Ib study of olaparib and carboplatin in BRCA1 or BRCA2 mutation-associated breast or ovarian cancer with biomarker analyses. J Natl Cancer Inst. 2014 May 19;106(6):dju089. doi: 10.1093/jnci/dju089. Print 2014 Jun. PMID 24842883
- [Background] O'Sullivan CC, Moon DH, Kohn EC, Lee JM. Beyond Breast and Ovarian Cancers: PARP Inhibitors for BRCA Mutation-Associated and BRCA-Like Solid Tumors. Front Oncol. 2014 Feb 28;4:42. doi: 10.3389/fonc.2014.00042. eCollection 2014. PMID 24616882
- [Background] Lee JM, Ledermann JA, Kohn EC. PARP Inhibitors for BRCA1/2 mutation-associated and BRCA-like malignancies. Ann Oncol. 2014 Jan;25(1):32-40. doi: 10.1093/annonc/mdt384. Epub 2013 Nov 12. PMID 24225019
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0050.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Ovarian Cancer Patients: Ovarian cancer patients with germline breast cancer mutation (gBRCAm) who have progressed on prior poly (ADP-ribose) polymerase inhibitor (PARPi) therapy BMN 673 (talazoparib): 1 mg by mouth (p.o.) once daily on 28-day cycles until disease progression
Period: Overall Study
Arm/Group | Ovarian Cancer Patients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ovarian Cancer Patients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (3.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Response (CR) + Partial Response (PR))
Description: Objective response (complete response (CR) + partial response (PR)) was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every 2 cycles, an average of 64 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer Patients
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the number participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events v4.0. For a detailed list of events, see the adverse event module.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ovarian Cancer Patients
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Duration of Response
Description: Duration of response is the time between study enrollment and off-treatment date.
Time Frame: 3 months
Measure: Median (Full Range); unit: months
Arm/Group | Ovarian Cancer Patients
Number analyzed (Participants) | 3
months | 2 [1 to 3]

4. Secondary Outcome: Progression Free Survival (PFS) on BMN673 (Talazoparib) to PFS From First Poly (ADP-ribose) Polymerase Inhibitor (PARPPi) Exposure
Description: The median time to progression after receiving BMN673 will be compared informally to the time of progression for the same patients after receiving an initial PARPi exposure. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more lesions is also considered progressions).
Time Frame: 3 months
Population: This outcome measure was not done because the study was prematurely closed by the Cancer Therapy Evaluation Program (CTEP) sponsor following the enrollment of 3 subjects. We were unable to analyze biomarker endpoints due to insufficient number of samples after premature closure of the study.
Arm/Group | Ovarian Cancer Patients
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Forkhead Box 03 (FOXO3a), p53-binding Protein 1 (53BP1) and RAD51 (i.e., Eukaryote Gene) Biomarkers
Description: Patients will undergo a mandatory biopsy at baseline and reverse phase protein microarray (RPPA)26 testing will be performed to determine the potential predictive biomarkers of subsequent poly (adenosine diphosphate [ADP]) ribose polymerase inhibitors (PARPi ) response.
Time Frame: Baseline
Population: Data was collected but was not analyzed given lack of statistical value of using only 3 samples and no follow up data.
Arm/Group | Ovarian Cancer Patients
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Secondary Mutation of Breast Cancer 1 (BRCA1) and Breast Cancer 2 (BRCA2)
Description: Patients will undergo a mandatory biopsy at baseline and Next Generation Sequencing to elucidate the secondary mutations of BRCA1 and BRCA2 will be performed.
Time Frame: Baseline
Population: Data was collected but was not analyzed given lack of statistical value of using only 3 samples and no follow up data.
Arm/Group | Ovarian Cancer Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Ovarian Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ovarian Cancer Patients (N=3)
Platelet Count Decreased (Investigations) | 1 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ovarian Cancer Patients (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (6)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Hyperhidrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (5)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vascular disorders - Other, bleeding gums (Vascular disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT02326844/Prot_SAP_ICF_000.pdf